CLINICAL TRIAL: NCT03757221
Title: A Multicentre Open-label Phase II Study of Ixazomib -Daratumumab Without Dexamethasone (IDara) in Elderly Relapse Refractory Multiple Myeloma
Brief Title: Ixazomib -Daratumumab Without Dexamethasone (IDara) in Elderly Relapse Refractory Multiple Myeloma
Acronym: IDARA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-070
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2018-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; daratumumab

STUDY DESIGN:
Intervention Model Description: We plan a single-arm non-randomized open label phase II study with a Fleming one stage hypothesis testing for the primary endpoint of VGPR (Very Good Partial Response) + CR (Complete Response) Rate during the twelve months follow-up. The efficacy of Daratumumab plus Ixazomib will be evaluated in comparison to a minimally effective lower threshold level of VGPR + CR.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination ixazomib + daratumumab without dexamethasone (Experimental): Elderly Relapse Refractory Multiple Myeloma Patients treated by Combination ixazomib + daratumumab without dexamethasone
  Interventions: Combination Product: Ixazomib and Daratumumab

INTERVENTIONS:
Combination Product: Ixazomib and Daratumumab — Daratumumab will be administrated every week for the first 2 cycles. For cycle 3 to 6, it will be administrated every two weeks at day 1 and day 15. From cycle 7 until progression Daratumumab will be administrated every 4 weeks.
  Ixazomib will be administrated every week three weeks on one week off at D1, D8 and D15 on a 28-d cycle basis.
  Dexamethasone will not be given except one series of 4 days of dexamethasone, 20 mg/day or a maximum of 80 mg, for emergencies and complications at initiation of treatment.

SUMMARY:
Multiple myeloma is an incurable hematological malignancy that affects older patients. Currently, despite recent progress, the disease relapses more or less quickly after initial treatment and requires the resumption of treatment with new drugs associated with cortisone, whose side effects are important. The investigators propose to conduct a phase 2 testing the combination ixazomib - daratumumab without dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to understand and voluntarily sign an informed consent form
* Must be able to adhere to the study visit schedule and other protocol requirements
* Age >= 65 years
* Subjects affiliated with an appropriate social security system.
* Life expectancy > 6 months
* Patients must have relapsed myeloma, and have been previously treated with Bortezomib, Melphalan and Prednisone (VMP) or Lenalidomide and Dexamethasone (Rd), or both:

  * One or two line(s) of prior therapies
  * Patients must have Progressive Disease as defined by the IMWG as one of the following (Kumar, 2016): Increase of 25% from lowest response value in any one or more of the following:

    * Serum M-component (absolute increase must be ≥ 0.5 g/100 ml) and/or Urine M-component (absolute increase must be ≥ 200 mg per 24 h) and/or
    * Only in patients without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels (absolute increase must be > 10 mg/l).
    * Bone marrow plasma cell percentage (absolute % must be ≥ 10%)
    * Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas
    * Development of hypercalcemia (corrected serum calcium > 11.5 mg/100 ml) that can be attributed solely to the plasma cell proliferative disorder
  * Patients must have undergone prior treatment with VMP or Rd:

    * They must have received at least two cycles of therapy
    * Either at diagnosis or relapse
* Patients must have a clearly detectable and quantifiable monoclonal M-component value: IgG (serum M-component > 10g/l) ; IgA (serum M-component > 5g/l) ; IgD (serum M-component > 0.5g/l); Light chain (serum M-component >1g/l or Bence Jones > 200 mg/24H) In patients without measurable serum and urine M-protein levels when the absolute serum Free Light chain (sFLC) is ≥100 mg/l and an abnormal sFLC K/λ ratio (<0.26 and >1.65) is found (Dispenzieri, 2008).
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Adequate bone marrow function within 5 days prior to 1st drug intake (cycle1, day 1, C1D1), without transfusion nor growth factor support within 5 days prior to 1st drug intake, defined as: Absolute neutrophils ≥ 1000/mm3 ; Platelets ≥ 50000/mm3 ; Haemoglobin ≥ 8.5g/dl
* Adequate organ function defined as: Serum creatinine clearance (MDRD formula) ≥30 ml/min ; Serum SGOT or SGPT < 3.0 X upper limit of normal (ULN) ; Serum total bilirubin < 1.5 ULN
* Wash out period of at least 2 weeks from previous antitumor therapy or any investigational treatment or 5 half-lives from previous antibodies.
* Women who are partners of men and of childbearing potential must be practicing one of the following methods of birth control: subcutaneous hormonal implant, levonorgestrel releasing intra-uterine system, medroxyprogesterone acetate depot, tubal sterilization, ovulation inhibitory progesterone only pills, or sexual intercourse with a vasectomized male partner (vasectomy must be confirmed by 2 negative semen analyses). Or women will commit to absolute and continuous abstinence confirmed to her physician on a monthly basis. Childbearing potential*. Contraception will start during therapy including dose interruptions, for 4 months after discontinuation of Ixazomib and Daratumumab.

Criteria for women of childbearing potential:

This protocol defines a female of childbearing potential as a sexually mature woman who:

1. has not undergone a hysterectomy or bilateral oophorectomy or
2. has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months)

   * A woman of childbearing potential must have 2 negative serum or urine pregnancy tests at Screening, first within 28 days prior to dosing and the second within 48 hours prior to dosing, and remain on a highly effective method of birth control. The two methods of reliable contraception must include one highly effective method and one additional effective (barrier) method. FCBP must be referred to a qualified provider of contraceptive methods if needed. The following are examples of highly effective and additional effective methods of contraception:

     * Highly effective methods: Intrauterine device (IUD) ; Hormonal (birth control pills, injections, implants) ; Tubal ligation ; Partner's vasectomy
     * Additional effective methods: Male condom ; Diaphragm CervicalCap
   * Serum (urine in the case where serum is not possible in a timely manner) pregnancy test to be performed for all women of childbearing potential regularly during the study, In addition, a pregnancy test may be done at any time during the study at the discretion of the investigator if a subject misses a period or has unusual menstrual bleeding.
   * A woman of childbearing potential must remain on a highly effective method of birth control. Contraception must begin 4 weeks before initiating treatment with Ixazomib and Daratumumab, during therapy, during dose interruptions and continuing for 4 months following discontinuation of Ixazomib and Daratumumab. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy.
   * A man who has not had a vasectomy and who is sexually active with a woman of childbearing potential must agree to use a barrier method of birth control eg, condom with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study, for 4 months following discontinuation of Ixazomib and Daratumumab. The exception to this restriction is that if the subject's female partner is surgically sterile, a second method of birth control is not required.

Exclusion Criteria:

* Target disease exceptions: Solitary bone/solitary extramedullary plasmocytoma ; Patients with non-secretory MM and non-measurable MM ; Evidence of central nervous system (CNS) involvement
* Medical history and Concurrent disease:

  * Subjects with prior (≤ 5 years) or concurrent invasive malignancies except the following: Adequately treated basal cell or squamous cell skin cancer ; Incidental finding of low grade (Gleason 3+3 or less) prostate cancer ; Any cancer from which the subject has been disease free for at least 3 years.
  * Subject with known/underlying medical conditions that, in the investigator's opinion would make the administration of the study drug hazardous (ie: uncontrolled diabetes or uncontrolled coronary artery disease)
  * Any uncontrolled or severe cardiovascular or pulmonary disease determined by the investigator including: NYHA functional classification III or IV congestive heart failure LVEF (Left Ventricular Ejection Fraction) ≥45% ; Uncontrolled angina, hypertension or arrhythmia Myocardial infarction in the past 6 months
  * Subjects with grade 2 or greater peripheral neuropathy (as per NCI-CTCAEv4.0)
  * Subject is a woman who is pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 4 months after the last dose of any component of the treatment regimen. Or, subject is a man who plans to father a child while enrolled in this study or within 4 months after the last dose of any component of the treatment regimen.
  * Known positive for HIV or active hepatitis B or C.
  * Subjects with psychiatric illnesses or social situations that would preclude them understanding the informed consent, study compliance or the ability to tolerate study procedures and/or study therapy
  * Subjects with known chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) < 50% of predicted normal. Note that FEV1 testing is required for patients suspected of having COPD and subjects must be excluded if FEV1 <50% of predicted normal.
  * Subjects with a history of moderate or severe persistent asthma within the past 2 years (see appendix), or with uncontrolled asthma of any classification at the time of screening (Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study).
  * Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of Ixazomib including difficulty swallowing.
* Physical and laboratory test findings:

  * Patients on dialysis or with a Creatinine clearance < 30mL/min
  * SGOT or SGPT >3ULN
* Prohibited prior therapies

  * Prior local irradiation within two weeks before first dose
  * Previous anti-CD38 therapy.
  * Previous Ixazomib therapy
* Allergies and Adverse Drug Reaction:Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Refusal to consent or protected by a legal regime (guardianship, trusteeship)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-02-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Very Good Partial Response (VGPR) + Complete Response (CR) Rate using the IMWG response criteria | 12 months
  The primary endpoint is the Very Good Partial Response (VGPR) + Complete Response (CR) Rate using the IMWG response criteria. Using IMWG criteria for best response reached at during the twelve months follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU CAEN Dept of Hematology, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided